CLINICAL TRIAL: NCT03060785
Title: Finding the Right Tenofovir/Emtricitabine Regimen for Pre-Exposure Prophylaxis (PrEP) in Transgender Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00092121
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: HIV Prevention
MeSH Terms: interventions — Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TFV/FTC dosing in Transgender women (Experimental): Single daily dose of oral Tenofovir Disoproxil Fumarate/Emtricitabine (Truvada)for 7days in transgender women taking feminizing hormones
  Interventions: Drug: Tenofovir Disoproxil Fumarate/Emtricitabine
- TFV/FTC dosing in Cis men (Active Comparator): Single daily dose of oral Tenofovir Disoproxil Fumarate/Emtricitabine (Truvada) for 7days in cis men
  Interventions: Drug: Tenofovir Disoproxil Fumarate/Emtricitabine

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate/Emtricitabine
  Other Names: Truvada

SUMMARY:
This is an open-label, steady-state study of Tenofovir (TFV) and Emtricitabine (FTC) pharmacokinetics (PK) in transgender women taking feminizing hormones. Half of the participants will be transgender women on feminizing hormones, the other half will be male volunteers not taking any hormone therapy.

DETAILED DESCRIPTION:
The investigators propose an open-label, steady-state study of TFV and FTC PK in blood and colon tissue in healthy TGW on feminizing hormones to be compared to healthy cis men, all at risk for HIV infection. Research participants will already have received eight days of TDF/FTC dosing. Evaluating TDF and FTC PK at steady-state is important as it reduces inter-individual variability since the rate of phosphorylation of TFV and FTC is highly variable, resulting in highly variable TFV-DP and Emtricitabine-Triphosphate (FTC-TP) PK among individuals in the first day and during rise to steady-state.

ELIGIBILITY:
Inclusion Criteria:

* TGW and cis men (male at birth and not a TGW)
* 18 to 65 years of age, inclusive on the date of screening
* Provides informed consent for the study
* Non-reactive HIV test results within four weeks of enrollment
* An estimated calculated creatinine clearance (eCcr) of at least 70 mL/min
* Agrees to use condoms for all sexual events during study participation.
* Taking daily oral Truvada® (Tenofovir disoproxil fumarate (TDF) 300 mg/Emtricitabine (FTC) 200 mg) for at least one week at the time of study PK sampling visit
* TGW have to be on an estradiol and have a serum total estradiol level > 100 picograms(pg)/ml

Exclusion Criteria:

* Significant colorectal symptom(s) as determined by medical history or by participant self-report
* Participant-reported symptoms and/or clinical or laboratory diagnosis of active rectal infection requiring treatment per current Centers for Disease Control (CDC) guidelines
* A positive test for Herpes Simplex Virus -2 (HSV-2) (individuals with active lesions only)
* Co-enrollment in any other HIV interventional research study (excluding behavioral only interventions) or prior enrollment in the active arm of a HIV vaccine trial.
* Positive hepatitis B surface antigen (HBsAg) test
* Interleukin therapy; medications with significant nephrotoxic potential, including but not limited to amphotericin B, aminoglycosides, cidofovir, foscarnet and systemic chemotherapy; medications that may inhibit or compete for elimination via active renal tubular secretion (including but not limited to probenecid); systemic immunomodulatory medications
* Participants with a history of having a gastrectomy, colostomy, ileostomy, or any other procedure altering the gastrointestinal tract or drug absorption
* Medications that prolong clotting time
* Any other condition or prior therapy that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, make the individual unsuitable for the study or unable to comply with the study requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender women (TGW) Cis men (male at birth and not a TGW)
Enrollment: 16 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Colon tissue tenofovir diphosphate (TFV-DP) | One week
  Endoscopy will be performed to obtain colorectal tissue biopsies. 15 biopsies will be collected and processed to isolate mucosal mononuclear cells (MMC). TFV-DP will be measured and reported as femtomoles per million cells (fmole/10E6 cells).

SECONDARY OUTCOMES:
Ex vivo colon explant HIV challenge | One week
  Colorectal tissue biopsies will be collected and exposed ex vivo to HIV and kept in culture for 15 days. Every three days a sample of fluid bathing the tissue sample will be tested for HIV p24 antigen. Results will be reported as picograms of p24 per milliliter (pg/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hendrix, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University Drug Development Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shieh E, Marzinke MA, Fuchs EJ, Hamlin A, Bakshi R, Aung W, Breakey J, Poteat T, Brown T, Bumpus NN, Hendrix CW. Transgender women on oral HIV pre-exposure prophylaxis have significantly lower tenofovir and emtricitabine concentrations when also taking oestrogen when compared to cisgender men. J Int AIDS Soc. 2019 Nov;22(11):e25405. doi: 10.1002/jia2.25405. PMID 31692269